CLINICAL TRIAL: NCT02841163
Title: Evaluation of Disc Resorption in Lumbar and Cervical Intervertebral Disc Herniation Patients Receiving Integrative Korean Medicine Treatment
Brief Title: Disc Resorption in Lumbar and Cervical Disc Herniation Patients Receiving Integrative Korean Medicine Treatment
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2016-06
Record Dates: First submitted 2016-06-27; First posted 2016-07-22 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Intervertebral Disc Displacement; Cervical Intervertebral Disc Displacement
Keywords: Magnetic Resonance Imaging; Patient Satisfaction; Numeric Rating Scale
MeSH Terms: conditions — Intervertebral Disc Displacement; Patient Satisfaction | interventions — Phytotherapy; Acupuncture Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumbar/cervical disc herniation group: Lumbar and cervical intervertebral disc herniation patients are administered integrative Korean medicine treatment consisting of herbal medicine, acupuncture, pharmacopuncture, bee venom pharmacopuncture, and Chuna manipulation.
  Interventions: Drug: Herbal medicine; Procedure: Acupuncture; Procedure: Pharmacopuncture; Procedure: Bee venom pharmacopuncture; Procedure: Chuna manipulation

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine was administered 2-3 times daily in water-based decoction (120ml) and dried powder (2g) form (Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, Saposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycine max, Atractylodes japonica).
  Other Names: Traditional herbal medicine
Procedure: Acupuncture — Acupuncture treatment was administered 1-2 times daily using mainly proximal acupuncture points and Ah-shi points.
Procedure: Pharmacopuncture — Select herbal ingredients (Eucommia ulmoides cortex, Acanthopanax sessiliflorum cortex, Achyranthis bidentata radix, Saposhnikovia divaricata radix, Cibotium barometz rhizoma, Paeonia albiflora radix alba, Ostericum koreanum radix, Angelica pubescens radix, and Scolopendra subspinipes corpus (Paeonia albiflora twice the proportion of that of other ingredients)) were freeze dried into powder form after decoction, then diluted in water-for-injection and adjusted for acidity and pH. Pharmacopuncture was administered once daily at Hyeopcheok (Huatuo Jiaji, EX B2), Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture was administered only after confirming a negative response to hypersensitivity skin tests. Diluted bee venom (saline:bee venom ratio, 10,000:1) filtered for allergens was injected at 4-5 acupoints proximal to the painful site at the physician's discretion. Each acupuncture point was injected to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
  Other Names: Bee venom acupuncture
Procedure: Chuna manipulation — Chuna is a Korean version of spinal manipulation that incorporates spinal manipulation techniques for mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manipulation was administered 3-5 times a week to pelvic, lumbar, thoracic, and cervical vertebrae at the physician's discretion.
  Other Names: Chuna spinal manipulation

SUMMARY:
Measurement of herniated disc resorption and assessment of satisfaction regarding post-treatment state and integrative Korean medicine treatment through phone interview in 500 patients with MRI follow-up results receiving treatment for lumbar and cervical disc herniation at Jaseng Hospital of Korean Medicine.

DETAILED DESCRIPTION:
Intervertebral disc herniation treatment can be largely divided into conservative and surgical approaches, and the greater majority of patients show relief of symptoms and resorption of herniated disc through non-surgical, conservative management. Despite concerns that early surgical interventions in intervertebral disc herniation without allowing for sufficient conservative treatment may indicate overtreatment, awareness and understanding in the general public is found somewhat lacking.

The objective of this study is to measure herniated disc resorption and assess satisfaction regarding post-treatment state and integrative Korean medicine treatment through phone interview in 500 patients with MRI follow-up results before and after receiving conservative treatment for lumbar and cervical disc herniation at Jaseng Hospital of Korean Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar and/or cervical disc herniation patients with baseline MRI and follow-up results after receiving treatment at Jaseng Hospital of Korean Medicine visiting between February 2012 and December 2015.
* Participants giving informed written consent to use of medical records for academic means.

Exclusion Criteria:

* Participants refusing to participate in study or to respond to phone interview.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lumbar and/or cervical disc herniation patients with MRI results before and after receiving treatment at Jaseng Hospital of Korean Medicine between February 2012 and December 2015
Sampling Method: Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Area of disc herniation at disc level most relevant to patient symptoms on MR sagittal and axial view | Change from baseline MRI (taken before treatment) at post-treatment completion MRI at average of 9 months
  Comparison of disc herniation in MRI between the baseline and post-treatment.

SECONDARY OUTCOMES:
Level of disc degeneration at disc level most relevant to patient symptoms on MR sagittal and axial view | Change from baseline MRI (taken before treatment) at post-treatment completion MRI at average of 9 months
  Level of disc degeneration at disc level most relevant to patient symptoms on MR sagittal and axial view will be classified into 5 levels according to the method suggested by Pfirrmann et al.
Level of disc herniation at disc level most relevant to patient symptoms on MR sagittal and axial view | Change from baseline MRI (taken before treatment) at post-treatment completion MRI at average of 9 months
  Level of disc herniation at disc level most relevant to patient symptoms on MR sagittal and axial view will be divided into 4 levels: protrusion, extrusion, sequestration, and migration
Level of herniated disc migration in patients with disc migration at disc level most relevant to patient symptoms on MR sagittal and axial view | Change from baseline MRI (taken before treatment) at post-treatment completion MRI at average of 9 months
  Level of herniated disc migration in patients with disc migration will be categorized into 3 levels in accordance with the Komori classification
Modic type change at vertebrae adjacent to disc level most relevant to patient symptoms on MR sagittal and axial view | Change from baseline MRI (taken before treatment) at post-treatment completion MRI at average of 9 months
  Modic type change at vertebrae adjacent to disc level most relevant to patient symptoms on MR sagittal and axial view will be classified into Modic types 0, 1, 2, and 3
Modic type change location with regard to disc level most relevant to patient symptoms on MR sagittal and axial view | Change from baseline MRI (taken before treatment) at post-treatment completion MRI at average of 9 months
  Location of modic type change at the vertebrae adjacent to the herniated disc is classified by whether it is above, below, neither above nor below, or both above and below the disc level most relevant to patient symptoms on MR sagittal and axial view
Pain NRS at site of chief complaint | Change from baseline MRI (taken before treatment) at post-treatment follow-up phone interview at average of 3 years
  Low back pain NRS or neck pain NRS
Radiating pain NRS associated with site of chief complaint | Change from baseline MRI (taken before treatment) at post-treatment follow-up phone interview at average of 3 years
  Radiating leg pain NRS or radiating arm pain NRS
Whether or not patient has been recommended for surgery regarding pain at site of chief complaint | Post-treatment follow-up phone interview at average of 3 years
  Whether or not patient has been recommended for surgery regarding pain at site of chief complaint will be recorded dichotomously
Whether or not pain has recurred for 1 month or longer at site of chief complaint | Post-treatment follow-up phone interview at average of 3 years
  Whether or not low back pain, radiating leg pain, neck pain or radiating arm pain has recurred at site of chief complaint will be recorded dichotomously
Type of treatment received, if any, for pain recurrence for 1 month or longer at site of chief complaint | Post-treatment follow-up phone interview at average of 3 years
  Type of treatment received, if any, for pain recurrence at site of chief complaint out of Korean medicine treatment, conventional nonsurgical treatment, or surgery will be recorded
Whether or not patient was aware of possible spontaneous disc resorption at site of chief complaint at onset | Post-treatment follow-up phone interview at average of 3 years
  Whether or not patient is aware of possible spontaneous disc resorption at site of chief complaint will be recorded dichotomously
Type of treatment patient would recommend to others as primary care | Post-treatment follow-up phone interview at average of 3 years
  Type of treatment patient would recommend to others out of surgical and nonsurgical treatment will be recorded
Satisfaction with integrative Korean medicine treatment | Post-treatment follow-up phone interview at average of 3 years
  Satisfaction with integrative Korean medicine treatment will be recorded using a 5-point Likert scale: very dissatisfied, dissatisfied, slightly satisfied, satisfied, very satisfied
Korean medicine treatment method perceived to be most effective | Post-treatment follow-up phone interview at average of 3 years
  Korean medicine treatment method perceived to be most effective out of herbal medicine, pharmacopuncture/bee venom pharmacopuncture, acupuncture, and Chuna manipulation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Joowon Kim, KMD, M.Sc., Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Medical Foundation, Bucheon-si, Gyeonggi Province, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Kim J, Shin JS, Lee YJ, Kim MR, Jeong SY, Choi YJ, Yoon TK, Moon BH, Yoo SB, Hong J, Ha IH. Long-Term Course to Lumbar Disc Resorption Patients and Predictive Factors Associated with Disc Resorption. Evid Based Complement Alternat Med. 2017;2017:2147408. doi: 10.1155/2017/2147408. Epub 2017 Jul 9. PMID 28769985